CLINICAL TRIAL: NCT04334356
Title: Pilot Testing of a Mobile Web App to Mitigate Posttraumatic Stress Symptoms (PTSS) After Sexual Assault
Brief Title: Testing of a Mobile Web App to Decrease Posttraumatic Stress Symptoms in Women After Sexual Assault
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-3399
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Anxiety Sensitivity; Chronic Pain; Sexual Assault
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain

STUDY DESIGN:
Intervention Model Description: In this pilot study, all participants will receive the active web app intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App Intervention (Experimental): All participants will receive the web app for prevention of posttraumatic stress.
  Interventions: Behavioral: Mobile Web App

INTERVENTIONS:
Behavioral: Mobile Web App — App for preventing development of posttraumatic stress based on cognitive behavioral techniques.

SUMMARY:
Interventions are available to all adult women sexual assault survivors to reduce the risk of pregnancy and sexually transmitted infection, yet no interventions are provided to reduce posttraumatic stress. This pilot study tests the ability of a smartphone-based web app to prevent and reduce posttraumatic stress in women sexual assault survivors.

ELIGIBILITY:
Inclusion Criteria:

* Present for emergency care within 72 hours of sexual assault
* Receive a sexual assault nurse examiner (SANE) exam
* Alert and oriented

Exclusion Criteria:

* Unable to consent due to intoxication, serious injury preventing ability to hear, speak, or see to consent, or other causes
* Prisoners
* Pregnant women
* Women living with assailant who plan to continue living with assailant
* Women with fractures from the assault
* Admitted patients
* Women who do not have a smartphone with continuous service for the past 12 months
* Inability to read and speak English
* No mailing address
* SANE exam took place >72 hours ago
* Patient previously enrolled in the study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as female/woman
Enrollment: 25 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Change from Week 6 to Month 6 in PCL-5 Scores | change from six weeks and six months
  The Posttraumatic Stress Disorder (PTSD) Checklist (PCL-5) for Diagnostic and Statistical Manual-5 (DSM-5) is the gold standard measure of PTSD symptom severity. Range: 0-80. Higher scores indicate worse outcomes. The investigators will assess whether reductions in PTSD symptoms from six weeks to six months are associated with reductions in anxiety sensitivity from the initial visit to six months. Change trajectories and mean scores of PCL-5 scores will be assessed over the 6 months of study follow-up. These patterns will be compared to prior observational research conducted in the lab.
Change from Week 6 to Month 6 in PROMIS Anxiety Scores | change from six weeks, and six months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety measures self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms (racing heart, dizziness) over the past seven days. Each question has five response options ranging in value from one to five (1=never; 2=rarely; 3=sometimes; 4=often; 5=always). To find the total raw score, sum the values of the response to each question. The lowest raw score is 8; the highest raw score is 40. A higher score represents more of the concept being measured. The investigators will assess whether reductions in PROMIS symptoms from six weeks to six months are associated with reductions in anxiety sensitivity from the initial visit to six months. Change trajectories and mean scores of PROMIS scores will be assessed over the 6 months of study follow-up. These patterns will be compared to prior observational research conducted in the lab.
Change from Baseline to Week 6 in ASI Scores | change from Initial to six weeks
  Anxiety Sensitivity Index-3 (ASI) is a 16-item self-report questionnaire that assesses fear of anxiety sensations. Each item is scored on a 5-point Likert scale (0 to 4) with total score ranging from a minimum of 0 to a maximum of 64 (higher scores indicate greater fear of anxiety sensations). The investigators will assess patterns of ASI scores over the 6 months of study follow-up, specifically using t-tests to test for change from intake to six weeks and six months.
Change from Week 6 to Month 6 in PROMIS Depression Scores | change from six weeks, and six months
  The PROMIS Depression assesses self-reported negative mood (sadness, guilt), views of self (self-criticism), and social cognition (loneliness), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose) over the past seven days. Each question has five response options ranging in value from one to five (1=never; 2=rarely; 3=sometimes; 4=often; 5=always). To find the total score, sum the values of the response to each question. The lowest raw score is 8; the highest is 40. A higher score represents more of the concept being measured. The investigators will assess whether reductions in PROMIS symptoms from six weeks to six months are associated with reductions in anxiety sensitivity from the initial visit to six months. Change trajectories and mean scores of PROMIS scores will be assessed over the 6 months of study follow-up. These patterns will be compared to prior observational research conducted in the lab.
Change from Week 6 to Month 6 in Pain Related to Assault | change from six weeks, and six months
  Pain Severity Numeric Rating Scale and Regional Pain Scale. The pain numeric rating scale (Pain NRS) consists of an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate worse pain. Participants chose the number that best described the pain during the last week. The investigators will assess whether reductions in pain NRS from six weeks to six months are associated with reductions in anxiety sensitivity from the initial visit to six months. Change trajectories and mean scores of pain NRS scores will be assessed over the 6 months of study follow-up. These patterns will be compared to prior observational research conducted in the lab.

SECONDARY OUTCOMES:
Insomnia Severity Index Scores | one week, six weeks, six months
  The Insomnia Severity Index (ISI) is a 7-item self-report questionnaire that provides a measure of insomnia severity based on several indicators (e.g., difficulty falling asleep, satisfaction with sleep, degree of impairment with daytime functioning). It has adequate internal consistency and temporal stability, has been validated against sleep diary and polysomnography data and was sensitive to change in several insomnia treatment studies. The ISI scale range is: minimum = 0, maximum = 28. Lower is considered 'better sleep', while higher is considered 'worse sleep/more insomnia'. This will be assessed at one week, six weeks, and six months to determine whether reductions in ISI from six weeks to six months are associated with reductions in anxiety sensitivity from the initial visit to six months. Change trajectories and mean scores of ISI scores will be assessed over the 6 months of study follow-up. These patterns will be compared to prior observational research conducted in the lab.
Somatic Symptoms | one week, six weeks, six months
  A previously used questionnaire from the investigator's lab will be used to measure somatic symptoms. This measure is a 21-item self-report measure assessing various somatic symptoms (e.g., headaches, fatigue, feeling faint, stomach distress). Items are rated on a 0-10 point scale, with total scores ranging from 0 to 210. Higher scores indicate worse symptoms. This will be assessed at one week, six weeks, and six months. The investigators will assess whether reductions in somatic symptoms from six weeks to six months are associated with reductions in anxiety sensitivity from the initial visit to six months. Change trajectories and mean scores of somatic symptoms scores will be assessed over the 6 months of study follow-up. These patterns will be compared to prior observational research conducted in the lab.
Association between Change in General Health and Anxiety Sensitivity | one week, six weeks, six months
  PROMIS Global Health-Physical Health Component. The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being. It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. Higher scores represent poorer health status. This will be assessed at one week, six weeks, and six months. The investigators will assess whether reductions in PROMIS symptoms from six weeks to six months are associated with reductions in anxiety sensitivity from the initial visit to six months. Change trajectories and mean scores of PROMIS scores will be assessed over the 6 months of study follow-up. These patterns will be compared to prior observational research conducted in the lab.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Short, PhD, Principal Investigator — University of Nevada, Las Vegas; Samuel McLean, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UCHealth Memorial Central Hospital, Colorado Springs, Colorado
  - University of North Carolina at Chapel Hill, SANE Program, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared by reasonable request beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available 9 to 36 months following publication and will remain available for five years.
Access Criteria: The investigator who proposes to use the data has IRB, IEC, or REB approval, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Broderick JE, DeWitt EM, Rothrock N, Crane PK, Forrest CB. Advances in Patient-Reported Outcomes: The NIH PROMIS((R)) Measures. EGEMS (Wash DC). 2013 Aug 2;1(1):1015. doi: 10.13063/2327-9214.1015. eCollection 2013. PMID 25848562